CLINICAL TRIAL: NCT03341715
Title: Metabotropic Glutamate Receptor-5 (mGlur5) Effects on Reward-Related fMRI-BOLD Activation in FHP and FHN
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HHC-2017-0172
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Familial Alcoholism Vulnerability
MeSH Terms: interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mavoglurant (AFQ056) (Experimental): The investigators will use a single dose of the AFQ056 (200 mg) versus placebo in random assignment single-blind fashion, administered 2 hours prior to the MRI and other measures, in two separate experimental study visits.
  Interventions: Drug: Mavoglurant (AFQ056)
- Placebo (Placebo Comparator): The investigators will use a single dose of the AFQ056 (200 mg) versus placebo in random assignment single-blind fashion, administered 2 hours prior to the MRI and other measures, in two separate experimental study visits.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mavoglurant (AFQ056) — 2-100mg tablets of Mavoglurant will be administered on the morning of 1 of the 2 experimental days by an RN or the physician investigator.
  Arms: Mavoglurant (AFQ056)
Other: Placebo — Two matching tablets of placebo will be administered on the morning of 1 of the 2 experimental days by an RN or the physician investigator.
  Arms: Placebo

SUMMARY:
The purpose of this pilot study is to evaluate the role of Mavoglurant in clarifying the neurobiology of alcoholism risk. This is a 1-site, randomized, within subjects, counterbalanced double-blind study of a single dose (200mg) of Mavoglurant and placebo.

DETAILED DESCRIPTION:
This project explores the effects of 1 dose of AZQ056, an experimental non-competitive antagonist to metabotropic glutamate receptor-5 (mGlur5) developed by Novartis, in a double-blind, randomized, counterbalanced manner on alcoholism risk-relevant tasks.

Drug/placebo will be administered on 2 separate visits separated by 1 week. More specifically, this project examines 4 functional MRI tasks related to different aspects of reward and/or impulsivity-related behavior in different contexts, compares the underlying neural circuitry across tasks, and uses a pharmacologic probe of the glutamatergic system to examine N-methyl-D-Aspartate and Dopamine (NMDA/DA) interactions.

The combined measures provide the opportunity to advance our understanding of specific aspects of brain function related to familial alcoholism vulnerability in an already well characterized population as some members evolve into alcohol abuse. In addition, as well as conventional within-task analyses, functional network connectivity and allied approaches will be used to examine brain networks across the above tasks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be first screened toxicologically for drugs of abuse (and for women of childbearing age, pregnancy) by urine testing, any positive test results in exclusion.
* Participants will be able to understand the procedures as judged by their ability to clearly repeat back to the PI or his designee correctly, the purpose and content of the planned research, and willingly agree to participate.

Exclusion Criteria:

1. a diagnosis of DSM-IV psychiatric disorder
2. report of psychotic disorder in a 1º relative, auditory or visual impairment that interferes with test-taking
3. prenatal exposure to alcohol plus currently meeting criteria for features of fetal alcohol syndrome
4. not speaking English fluently or being a non-native English speaker, or being educated in a primary language other than English > grade 1
5. mental retardation (Full Scale IQ<70)
6. traumatic brain injury with loss of consciousness > 30 minutes or concussion in last 30 days
7. presence or history of any medical/neurologic illness that may affect brain physiology (e.g., epilepsy, Multiple Sclerosis), including focal brain lesion seen on structural MRI (all structural scans are read by a licensed radiologist)
8. current pregnancy (all females will be tested with urine screens on the day of MRI);
9. All participants will receive a urine screen for the presence of marijuana, cocaine, opiates and a breath screen to detect the presence of alcohol
10. Inability to comprehend the consent form appropriately
11. Other specific fMRI exclusions include metal devices, clips or fragments in body (orbital x-ray performed if needed).

    * Individuals will be excluded who have taken, within the prior 14 days, the following strong inhibitors or inducers of CYP1A, CYP2C, and CYP3A and CYP3A4: iprofloxacin, enoxacin, fluvoxamine; gemfibrozil; fluconazole, fluvoxamine, ticlopidine; boceprevir, clarithromycin, conivaptan, grapefruit juice, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, voriconazole; bupropion, fluoxetine, paroxetine, quinidine; avasimibe, carbamazepine, phenytoin, rifampin, and St. John's wort.
    * Individuals will also be excluded who have taken, within 14 days, the following moderate inhibitors and inducers of CYP3A: Amprenavir, aprepitant, atazanavir, ciprofloxacin, crizotinib, darunavir/ritonavir, diltiazem, erythromycin, fluconazole, fosamprenavir, imatinib, and verapamil; and bosentan, efavirenz, etravirine, modafinil, and nafcillin.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
MRI Monetary Incentive Delay (MID) task | 2 Hours post medication administration
  BOLD activation during A1 phase of MID

SECONDARY OUTCOMES:
MRI Alcohol Cue Reactivity (ACR) task | 2 Hours post medication administration
  BOLD signal activation in the fusiform area and hippocampus for the alcohol cue reactivity (ACR) task. FHP individuals will show increased BOLD signal activation in the fusiform area and hippocampus to repeated alcohol images.

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States